CLINICAL TRIAL: NCT04383106
Title: Bowel Colonization With Multi-drug Resistant Bacterial Species in Hospitalized Patients With acute-on Chronic Liver Failure (ACLF), and Its Relationship With Extra-intestinal Infectious Events and Short-term Outcomes.
Status: Completed | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: ILBS-ACLF-10
Record Dates: First submitted 2020-04-22; First posted 2020-05-12 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Acute-On-Chronic Liver Failure
MeSH Terms: conditions — Acute-On-Chronic Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Bowel colonization with anti-microbial resistant bacteria increases the risk of clinical infections. Infections caused by anti-microbial resistant bacteria have been associated with increased mortality, prolonged hospital stay, and increased costs. In addition, with the emergence of carbapenemase resistant bacterial species, there may not be any effective therapy for patients infected with such resistant species.

Bowel colonization with anti-microbial resistant bacteria is an established risk factor for infections due to resistant bacteria, especially in transplanted patients and in intensive care unit. In this study we will study whether bowel colonisation in Acute on Chronic Liver Failure patient increases the risk of infection development in extra intestinal sites.

ELIGIBILITY:
Inclusion Criteria:

- Patients with Acute on Chronic Liver Failure admitted to the ward/High Dependency Unit/Intensive Care Unit.

Exclusion Criteria:

1. Patients on immunosuppressant medications or on daily steroids (excluding inhaled steroids) or >2 weeks.
2. Patients with additional primary or acquired immunosuppressive states like hypogammaglobinemia, post-splenectomy, human immunodeficiency virus (HIV) infection etc.
3. Neutropenia defined as absolute neutrophil count or total white blood cell count (WBC) <500/mm3
4. Patients with extra-hepatic malignancy or on cytotoxic chemotherapy.
5. Patients with ileus, bowel hypomotility, severe constipation requiring laxatives/purgatives or enemas to evacuate.
6. Patients with fresh or altered blood in stools.
7. Patients with anatomical predisposition to infection/ bacterial seeing like prosthesis or foreign body. Patients with exfoliative skin conditions, significant mucosal ulcerations, or skin ulcers. Patients who have received > 2 weeks of antibiotics before current admission.
8. Pregnant patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: All patients admitted to the Institute of Liver and Biliary Sciences (ILBS) with Acute on Chronic Liver Failure (ACLF) will be evaluated for inclusion. ACLF will be defined by the Asian Pacific association for the Study of Liver Disease (APASL) criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Fecal isolation rates of carbapenem resistant gram negative bacterial species (CR-GNB) among hospitalized ACLF patients | Day 28

SECONDARY OUTCOMES:
Fecal isolation rates of Extended Spectrum Beta-Lactamases (ESBL) producing gram negative bacterial species among hospitalized ACLF patients. | Day 28
Fecal isolation rates of Vancomycin-resistant enterococci (VRE) species among hospitalized ACLF patients | Day 28
Fecal carriage rates of C. difficile among hospitalized ACLF patients. | Day 28
Correlation of fecal carriage of resistant bacterial species with antibiotic exposure antibiotic type and duration | Day 28
Concordance of bowel colonizing resistant bacterial species, with concurrent or subsequent infecting bacterial isolates from extra-intestinal sites | Day 28
  Stool culture sensitivity organism concordance will be checked with culture organism from other sites like blood, urine, ascitic, pleural, skin.
Factors predisposing patients colonized with resistant bacterial species to develop extra-intestinal infectious events due to the same species | Day 28
  Factors will be assessed like previous hospitalisation, days of hospital stay, severity of disease, number and type and dosage of antibiotics usage in previous hospitalisation and current hospital stay, other symptom localisation of extraintestinal sites like lung infection, abdominal infection, urine infection, skin infection
Timeline of bowel colonization with resistant bacterial species among hospitalized ACLF patients | Day 28
Correlation of the fecal carriage rates of resistant bacterial species with etiology and severity of ACLF, including onset and resolution of organ failure (OF). | Day 28
Correlation of fecal carriage resistant bacterial species with patient outcomes (admission duration or survival duration, short-term survival to discharge, readmission rates, and 30-day survival | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Singh SP, Bhatia V, Kale P, Kumar G, Khillan V, Vijayaraghavan R. Bowel Colonization With Carbapenem-Resistant Bacteria Is Associated With Short-Term Outcomes in Patients With Acute-On-Chronic Liver Failure. J Gastroenterol Hepatol. 2025 Feb;40(2):528-536. doi: 10.1111/jgh.16830. Epub 2024 Nov 20. PMID 39568042